CLINICAL TRIAL: NCT00093470
Title: A Phase III Randomized Study of Farnesyl Transferase Inhibitor R115777 in Acute Myeloid Leukemia (AML) Patients in Second or Subsequent Remission or in Remission After Primary Induction Failure or Patients Over Age 60 in First Remission
Brief Title: Tipifarnib in Treating Patients With Acute Myeloid Leukemia in Remission
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00535; NCI-2009-00535 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); E2902; E2902 (Other: ECOG-ACRIN Cancer Research Group); E2902 (Other: CTEP); U10CA180820 (NIH); U10CA021115 (NIH)
Record Dates: First submitted 2004-10-06; First posted 2004-10-08 (Estimated); Results first posted 2015-11-10 (Estimated); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Adult Acute Megakaryoblastic Leukemia; Adult Acute Monocytic Leukemia; Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With Inv(16)(p13.1q22); CBFB-MYH11; Adult Acute Myeloid Leukemia With Maturation; Adult Acute Myeloid Leukemia With Minimal Differentiation; Adult Acute Myeloid Leukemia With t(16;16)(p13.1;q22); CBFB-MYH11; Adult Acute Myeloid Leukemia With t(8;21); (q22; q22.1); RUNX1-RUNX1T1; Adult Acute Myeloid Leukemia With t(9;11)(p22.3;q23.3); MLLT3-KMT2A; Adult Acute Myeloid Leukemia Without Maturation; Adult Acute Myelomonocytic Leukemia; Adult Erythroleukemia; Adult Pure Erythroid Leukemia; Alkylating Agent-Related Acute Myeloid Leukemia; Myelodysplastic Syndrome With Excess Blasts; Recurrent Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Myeloid, Acute; Leukemia, Erythroblastic, Acute; Anemia, Refractory, with Excess of Blasts | interventions — Watchful Waiting; Observation; tipifarnib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (tipifarnib) (Experimental): Patients receive tipifarnib PO BID on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Tipifarnib
- Arm B (clinical observation) (Other): Patients undergo observation only.
  Interventions: Procedure: Clinical Observation

INTERVENTIONS:
Procedure: Clinical Observation — Undergo observation
  Other Names: observation
  Arms: Arm B (clinical observation)
Drug: Tipifarnib — Given PO
  Other Names: R115777; Zarnestra
  Arms: Arm A (tipifarnib)

SUMMARY:
This randomized phase III trial studies tipifarnib in treating patients with acute myeloid leukemia (AML) in remission. Tipifarnib may stop the growth of cancer cells by blocking the enzymes necessary for their growth. It is not yet known whether tipifarnib is more effective than observation alone in preventing the recurrence of AML.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare R115777 (tipifarnib) maintenance therapy to observation only with respect to disease-free survival (DFS) in patients with AML in second or subsequent complete remission or in complete response (CR) following primary induction failure.

SECONDARY OBJECTIVES:

I. To compare overall survival of patients in both arms. II. To evaluate the long-term safety and toxicity of extended administration of R115777 in AML patients in remission.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive tipifarnib orally (PO) twice daily (BID) on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM B: Patients undergo observation only.

After completion of study treatment, patients are followed up for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible to enter this study must fall into one of these categories:

  * Patients in first remission following primary induction failure
  * Patients must have received at least two chemotherapy induction regimens
  * Patients in second or subsequent remission
  * Patients > 60 years old in first remission
* Patients must be in complete remission (CR) or morphologic remission (MR) by blood counts and bone marrow studies to enter the study

  * Confirmatory bone marrow must be performed =< 2 weeks prior to randomization
* Patients must have morphologic proof (from bone marrow aspirate, smears or touch preps of marrow biopsy) that they had AML of one of the following types prior to achievement of CR/MR

  * Acute myeloblastic leukemia, minimal differentiation (French-American-British [FAB] M0)
  * Acute myeloblastic leukemia without differentiation (FAB M1)
  * Acute myeloblastic leukemia with maturation (FAB M2)
  * Acute myelomonocytic leukemia (FAB M4)
  * Acute monocytic leukemia (FAB M5)
  * Acute erythroleukemia (FAB M6)
  * Acute megakaryocytic leukemia (FAB M7)
  * Refractory anemia with excess blasts in transformation (RAEB-T)
  * AML by World Health Organization (WHO) criteria
  * Acute myeloid leukemia with multilineage dysplasia
* Patients with acute promyelocytic leukemia (FAB M3) are not eligible
* Patients must be registered within 60 days of completion of therapy for the current remission; patients are eligible if they meet any of the criteria below:

  * Within 60 days of remission (CR or MR) by peripheral blood counts following induction therapy or
  * Within 60 days of discharge from the hospital following induction therapy or
  * Within 60 days of discharge from the hospital following post-remission therapy or
  * Within 60 days of recovery of blood counts following last dose of chemotherapy
* All of the patients below are eligible for study entry:

  * Patients who have received consolidation therapy
  * Patients who have not received any consolidation or post remission therapy
  * Patients who have had an autologous stem cell transplant
* Patients who have received an allogeneic transplant (bone marrow transplant [BMT] or peripheral stem cell transplant [PSCT]) in their current remission are ineligible; patients who have had an allogeneic transplant in a previous remission and are currently in remission after subsequent relapse are eligible
* Patients with a history of extramedullary disease are eligible if they are in complete remission at the time of study entry and no longer requiring therapy for their extramedullary disease
* Patients must not be pregnant or breast-feeding; all females of childbearing potential must have a blood test or urine study < 2 weeks prior to randomization to rule out pregnancy
* Women of childbearing potential and sexually active males are strongly advised to use an accepted and effective method of contraception
* Patients must not be known to have an allergy to imidazole drugs, such as clotrimazole ketoconazole, miconazole, econazole, or terconazole; this does not include fluconazole, voriconazole, or itraconazole
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2
* Patients must not have active cardiac or pulmonary disease; but patient will be eligible if disease is medically controlled
* Patients must not have active renal disease; creatinine must be =< 1.5 x upper limit of normal
* Patients must not have active hepatic disease; total or direct bilirubin must be < 2 mg/dl
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) must be =< 2.5 times the upper limit of normal
* Absolute neutrophil count (ANC) >= 1000/mm^3
* Platelet count >= 50,000/mm^3
* Patients must not be taking a hepatic enzyme-inducing anti-convulsant; a patient will not be eligible for the study if the patient is currently taking one of these agents and cannot be switched to a non-hepatic enzyme-inducing anti-convulsant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2004-08-18 (Actual); Primary Completion 2015-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Selina Luger, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (341):
- United States (339):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program NCORP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Saint Francis Hospital - Wilmington, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hematology Oncology Associates of Eastern Idaho, Idaho Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Jesse Brown Veterans Affairs Medical Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Mercy Hospital and Medical Center, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Eureka Hospital, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Midwest Center for Hematology Oncology, Joliet, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - Deerpath Medical Associates, Lake Forest, Illinois
  - NorthShore Hematology Oncology-Libertyville, Libertyville, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Franciscan St. James Health-Olympia Fields Campus, Olympia Fields, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Sarah Culbertson Memorial Hospital, Rushville, Illinois
  - Edward H Kaplan MD and Associates, Skokie, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Midwest Cancer Research Group Incorporated, Skokie, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - The Community Hospital, Munster, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Heartland Oncology and Hematology LLP, Council Bluffs, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Genesis Medical Center - West Campus, Davenport, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Hospital District Sixth of Harper County, Anthony, Kansas
  - Memorial Hospital of Arkansas City, Arkansas City, Kansas
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Ottawa, Ottawa, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Shawnee Mission Medical Center-KCCC, Shawnee Mission, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Saint Francis Hospital and Medical Center - Topeka, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center/Terrebonne General Medical Center, Houma, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Overton Brooks Veteran's Administration Medical Center, Shreveport, Louisiana
  - Louisiana State University Health Sciences Center Shreveport, Shreveport, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine General Medical Center-Thayer, Waterville, Maine
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Franklin Medical Center, Greenfield, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Providence Hospital-Southfield Cancer Center, Southfield, Michigan
  - Medini, Eitan MD (UIA Investigator), Alexandria, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Etzell, Paul S MD (UIA Investigator), Fergus Falls, Minnesota
  - Swenson, Wade II, MD (UIA Investigator), Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Hattiesburg Clinic - Hematology/Oncology Clinic, Hattiesburg, Mississippi
  - Hematology and Oncology Clinic, Hattiesburg, Mississippi
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Deaconess Medical Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Internal Medicine of Bozeman, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Eastern Montana Cancer Center, Miles City, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Orange Regional Medical Center, Middletown, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center-Wakefield Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Akron General Medical Center, Akron, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - The Jewish Hospital, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Cancer Care Associates, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Mercy Hospital, Scranton, Pennsylvania
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - AnMed Health Hospital, Anderson, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Baylor Saint Luke's Medical Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Michael E DeBakey VA Medical Center, Houston, Texas
  - The Methodist Hospital System, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Cottonwood Hospital Medical Center, Murray, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Intermountain Health Care, Salt Lake City, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont College of Medicine, Burlington, Vermont
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Central Washington Hospital, Wenatchee, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Sacred Heart Hospital, Eau Claire, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Ascension Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - Saint Michael's Hospital, Stevens Point, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Welch Cancer Center, Sheridan, Wyoming
- Rambam Medical Center, Haifa, Israel
- Instituto Nacional de Enfermedades Neoplasicas, Lima, Peru

REFERENCES:
- See also: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on August 18, 2004, suspended between August 8, 2007 and February 6, 2008 for toxicity and safety evaluation, and closed on December 7, 2009 with a total of 144 patients accrued.
Period: Overall Study
Arm/Group | Arm A (Tipifarnib) | Arm B (Clinical Observation)
Started | 73 | 71
Treated | 72 | 71
Patients With Toxicity Assessment | 72 | 69
Completed | 0 (Treatment continued until disease progression or unacceptable toxicities.) | 71 (Patients underwent observation only.)
Not Completed | 73 | 0
Not completed — Disease progression | 39 | 0
Not completed — Adverse Event | 15 | 0
Not completed — Death | 2 | 0
Not completed — Withdrawal by Subject | 8 | 0
Not completed — Alternative therapy | 2 | 0
Not completed — Other complicating disease | 3 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Never started treatment | 1 | 0
Not completed — ANC < 1000 on day 1 of cycle 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Tipifarnib) | Arm B (Clinical Observation) | Total
Number analyzed (Participants) | 73 | 71 | 144
Age, Continuous [Median (Full Range); unit: years] | 70 [30 to 86] | 69 [28 to 80] | 69 [28 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 34 | 71
  Male | 36 | 37 | 73

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival
Description: Disease-free survival (DFS) is defined as the time from randomization to relapse or death without relapse.
Time Frame: Assessed monthly for the first 6 months then every 3 months or as clinically indicated, up to 5 years.
Population: All randomized patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Tipifarnib) | Arm B (Clinical Observation)
Number analyzed (Participants) | 73 | 71
months | 8.87 [5.85 to 13.34] | 5.26 [3.88 to 7.56]
Statistical Analysis 1: Comparison: Arm A (Tipifarnib) vs Arm B (Clinical Observation); Test type: Superiority or Other; p = 0.026, Log Rank — one-sided p-value; threshold for statistical significance <0.025; stratified log rank test; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.538 to 1.072] — Hazard ratio of DFS for Arm A to Arm B

2. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined as the time from randomization to death from any cause.
Time Frame: Assessed monthly for the first 6 months then every 3 months or as clinically indicated, up to 5 years.
Population: All randomized patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Tipifarnib) | Arm B (Clinical Observation)
Number analyzed (Participants) | 73 | 71
months | 16.36 [12.26 to 25.20] | 9.27 [8.41 to 19.88]
Statistical Analysis 1: Comparison: Arm A (Tipifarnib) vs Arm B (Clinical Observation); Test type: Superiority or Other; p = 0.056, Log Rank — one-sided p-value; threshold for statistical significance < 0.025; stratified log rank test; Hazard Ratio (HR) = 0.809, 95% CI 2-sided [0.567 to 1.155] — Hazard ratio of OS for Arm A to Arm B

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment
Arm/Group | Arm A (Tipifarnib) | Arm B (Clinical Observation)
Serious Adverse Events (participants affected / at risk) | 52/72 | 8/69
Other Adverse Events (participants affected / at risk) | 50/72 | 23/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Tipifarnib) (N=72) | Arm B (Clinical Observation) (N=69)
Anemia (Blood and lymphatic system disorders) | 9 | 2
White blood cell decreased (Investigations) | 29 | 2
Neutrophil count decreased (Investigations) | 25 | 0
Platelet count decreased (Investigations) | 36 | 6
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0
Catheter related infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Peripheral nerve infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
GGT increased (Investigations) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Confusion (Psychiatric disorders) | 2 | 0
Agitation (Psychiatric disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Psychosis (Psychiatric disorders) | 1 | 0
Eye disorders - Other, specify (Eye disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Tipifarnib) (N=72) | Arm B (Clinical Observation) (N=69)
Anemia (Blood and lymphatic system disorders) | 40 | 13
White blood cell decreased (Investigations) | 42 | 12
Neutrophil count decreased (Investigations) | 4 | 0
Platelet count decreased (Investigations) | 39 | 11
Fatigue (General disorders) | 5 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less